CLINICAL TRIAL: NCT02810912
Title: Gastroesophageal Regurgitation During Perioperative Period Under General Anesthesia: a Pilot Study With Multichannel Intraluminal Impedance-pH Monitoring
Brief Title: Gastroesophageal Regurgitation Under General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201603012RIND
Record Dates: First submitted 2016-06-12; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: The Episodes of Gastric Regurgitation
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Supraglottic airway device-based anesthesia: Investigators planned to enroll 200 cases who will receive scheduled surgery under supraglottic airway device-based general anesthesia.
  Interventions: Other: the effect of surgical position

INTERVENTIONS:
Other: the effect of surgical position — Investigators do not have intervention in the observation study. Investigators only use the MII-pH catheter to observe the episodes of gastric regurgitation in patients receiving supraglottic airway device under general anesthesia. Thus, investigators are going to observe the effect of surgical position change, body weight, surgical time. And investigators will have a control group, which patients undergo elective surgeries without surgical position change, no longer surgical time, and normal range of body weight.
  Other Names: the effect of body weight; The effect of surgical time; The standard elective surgery as control group

SUMMARY:
Gastric regurgitation increases the risk of pulmonary aspiration in surgical patients receiving general anesthesia because of depression of gastro-esophageal reflux. In addition, some patients may have higher risk of aspiration as a result of reduced gastric emptying and gastroesophageal reflux, prolonged surgical time, and laparoscopic surgery. Second-generation supraglottic airway device (SAD) provides an additional channel to facilitate the drainage the gastric content to prevent from aspiration, which was routinely used in surgeries. Currently, multichannel intraluminal impedance-pH (MII-pH) monitoring, which combines multiple impedance channels to conventional pH catheters, is regarded as the most sensitive technique for detecting reflux events. Therefore, application of MII-pH monitoring on the SAD-based general anesthesia may help to detect ongoing reflux/regurgitation in the esophagus of patients during perioperative period. The hypothesis of the present study is that the occurrences of gastroesophageal regurgitation during general anesthesia may be influenced by the several factors, such as abdominal insufflation during laparoscopy, longer surgical time, Trendelenburg position, higher body weight, etc.

DETAILED DESCRIPTION:
Investigators aim to observe the occurrences of gastroesophageal regurgitation through the continuous monitoring with the novel technique of MII-pH during the perioperative period of a variety of common surgical procedures under SAD-based general anesthesia in this pilot study. Furthermore, investigators will also determine the factors associated with the occurrence of gastroesophageal regurgitation during these various surgical procedures under general anesthesia.

Investigators include the patients who will receive scheduled surgery under SAD-based general anesthesia and aged >= 20 will be enrolled. All subjects provide basic demographic data and fill in standard symptom questionnaire for evaluation of baseline severity of gastroesophageal reflux and other associated gastrointestinal and sleep symptoms. Supraglottic airway device with i-gel will be inserted to establish airway, and the gastric content will be suctioned out through the esophageal vent of i-gel. MII-pH catheter will be inserted though the esophageal vent of i-gel to detect and characterize gastroesophageal reflux events in the perioperative period. After removal of SAD, the patients were follow the saturation, sore throat or hoarseness in the postoperative care unit, as well as the possible complications.

Investigators will not only elucidate the clinical characteristics and risk factors in patients receiving elective surgeries, but also determine the severity of gastric regurgitation during the intraoperative period.

Investigators will correlate the reflux pattern, frequency, content and proximal extent of all reflux events and symptom correlation with clinical features in the intraoperative period. The study results could help us study more in the gastric regurgitation in perioperative period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will receive scheduled surgery under SAD-based general anesthesia
2. Aged >= 20

Exclusion Criteria:

1. Major systemic disease, such as congestive heart failure, liver cirrhosis, end stage renal disease and malignancy.
2. Patients who have the risk of difficult ventilation or intubation.
3. pregnant women
4. prior nasal surgery or trauma
5. current use anticoagulant or antiplatelet agents
6. coagulopathy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who will receive scheduled surgery under supraglottic airway device-based general anesthesia and aged >= 20 will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-06; Primary Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
episode of gastric regurgitation | From the insertion of supraglottic airway device until removal of supraglottic airway device, whichever came first, assessed up to the total anesthetic time.
  MII-pH catheter will be inserted though the esophageal vent of i-gel to detect and characterize gastroesophageal reflux during the perioperative period. Continuous recording will be performed for perioperative period to assess the severity of gastric regurgitation. The data will be analyzed using the package analysis software and will then be reviewed by software and corrected manually by an experienced gastroenterologist. Reflux numbers and reflux type (liquid and mixed), acidic (acid, weak-acid, alkaline) and proximal extent (height above LES) will be determined.
  The definition of total anesthetic time is from induction to removal of the i-gel.

SECONDARY OUTCOMES:
the effect of surgical position in episode of gastric regurgitation | From the insertion of supraglottic airway device until removal of supraglottic airway device, whichever came first, assessed up to the total anesthetic time.
  MII-pH catheter will be inserted though the esophageal vent of i-gel to detect and characterize gastroesophageal reflux during the perioperative period. Continuous recording will be performed for perioperative period to assess the severity of gastric regurgitation. The investigators aim to observe the effect of surgical position in episode of gastric regurgitation. The data will be analyzed using the package analysis software and will then be reviewed by software and corrected manually by an experienced gastroenterologist. Reflux numbers and reflux type (liquid and mixed), acidic (acid, weak-acid, alkaline) and proximal extent (height above LES) will be determined.

OTHER OUTCOMES:
the effect of body weight in episode of gastric regurgitation | From the insertion of supraglottic airway device until removal of supraglottic airway device, whichever came first, assessed up to the total anesthetic time.
  MII-pH catheter will be inserted though the esophageal vent of i-gel to detect and characterize gastroesophageal reflux during the perioperative period. Continuous recording will be performed for perioperative period to assess the severity of gastric regurgitation. The investigators aim to observe the effect of body weight (BMI in kg/m2, weight in kilograms,height in meters) in episode of gastric regurgitation. The data will be analyzed using the package analysis software and will then be reviewed by software and corrected manually by an experienced gastroenterologist. Reflux numbers and reflux type (liquid and mixed), acidic (acid, weak-acid, alkaline) and proximal extent (height above LES) will be determined.
The effect of anesthetic time in episode of gastric regurgitation | From the insertion of supraglottic airway device until removal of supraglottic airway device, whichever came first, assessed up to the total anesthetic time.
  MII-pH catheter will be inserted though the esophageal vent of i-gel to detect and characterize gastroesophageal reflux during the perioperative period. Continuous recording will be performed for perioperative period to assess the severity of gastric regurgitation. The investigators aim to observe the effect of surgical time in episode of gastric regurgitation. The data will be analyzed using the package analysis software and will then be reviewed by software and corrected manually by an experienced gastroenterologist. Reflux numbers and reflux type (liquid and mixed), acidic (acid, weak-acid, alkaline) and proximal extent (height above LES) will be determined.

IPD SHARING:
Plan to Share IPD: No
We did not plan to share our data, because it involved the patients' privacy.